CLINICAL TRIAL: NCT02163096
Title: A Study to Assess Benign Joint Hypermobility Syndrome in Children With a History of Wheezing or Asthma
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Ronald L. Morton, Professor of Pediatrics, University of Louisville
Other Study IDs: 14.0447
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Benign Joint Hypermobility Syndrome; Wheezing; Asthma
MeSH Terms: conditions — Respiratory Sounds; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- History of Wheezing, Benign Joint Hypermobility Syndrome
- Asthma, Benign Joint Hypermobility Syndrome

SUMMARY:
The purpose of this study is to assess benign joint hypermobility syndrome (BJHS) in children with a history of wheezing or asthma. BJHS is a common syndrome of joint and connective tissue laxity without any other rheumatologic disease. This assessment will be performed by using either method below depending upon if the child has a history of wheezing or severe asthma:

1. Determine the correlation, if there is an increased rate of BJHS in children with a history of wheezing as well as if there is an increased history of wheezing in children with BJHS; or
2. Determine asthma control, lung function and asthma exacerbations (a flare up or acute worsening of symptoms) in children with BJHS compared to children with asthma without BJHS, to assess if it BJHS is associated more with children with severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* All children ages 6-16 with a history of wheezing or asthma

Exclusion Criteria:

* For subjects with a history of Wheezing: History of chronic lung disease or prematurity, chronic aspiration, congenital anomalies of the upper and lower airway, primary ciliary dyskinesia, cystic fibrosis, history of heart failure, immune deficiency, or any inflammatory arthritis.
* For Subjects with a history of Asthma: current acute respiratory exacerbation, history of chronic lung disease of prematurity, chronic aspiration, congenital anomalies of the upper or lower airway, primary ciliary dyskinesia, cystic fibrosis, restrictive lung disease, history of heart failure, immune deficiency, or inflammatory arthritis.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 6-16 in Primary Care Clinic and Pediatric Subspecialty Clinics of Pulmonary and Allergy/Immunology.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determine correlation between BJHS and Wheezing/Asthma | 6 months
  Determine the correlation, if there is an increased rate of BJHS in children with a history of wheezing as well as if there is an increased history of wheezing in children with BJHS, enrolled during well child visits and perform physical exams to screen for BJHS using a standardized assessment, Beighton Criteria, where a score is reached by testing the range of motion of the child's joints to determine if they are more loose than normal.
  Pediatric asthma patients will participate by, either the caregiver or child filling out a questionnaire to assess asthma control and history of exacerbation. Spirometry, a pulmonary lung function test, will be performed on all subjects along with a physical exam to screen for BJHS using standardized assessment, Beighton Criteria, where a score is reached by testing the range of motion of the child's joints to determine if they are more loose than normal.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Louisville - Sam Swope Kosair Charities Centre, Louisville, Kentucky
  - University of Louisville Allergy and Immunology, Louisville, Kentucky
  - University of Louisville Pediatric Pulmonology, Louisville, Kentucky